CLINICAL TRIAL: NCT01426126
Title: Phase II Study of Genexol-PM, a Cremophor-free, Polymeric Micelle Formulation of Paclitaxel for Patients With Advanced Urothelial Cancer Previously Treated With Gemcitabine and Platinum
Brief Title: Study of Genexol-PM in Patients With Advanced Urothelial Cancer Previously Treated With Gemcitabine and Platinum
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Samsung Medical Center (Other); Kangdong Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Jin-Hee Ahn, Associate professor, Asan Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UOSG-AMC-0702
Record Dates: First submitted 2011-08-29; First posted 2011-08-31 (Estimated); Last update posted 2011-12-07 (Estimated); Status verified 2011-12

CONDITIONS: Bladder Cancer; Ureter Cancer
Keywords: urothelial carcinoma; gemcitabine; platinum; refractory; salvage chemotherapy
MeSH Terms: conditions — Urinary Bladder Neoplasms; Ureteral Neoplasms; Carcinoma, Transitional Cell | interventions — genexol-PM

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Genexol PM (Experimental): Genexol PM intravenous infusion every 3 weeks
  Interventions: Drug: Genexol PM

INTERVENTIONS:
Drug: Genexol PM — Genexol-PM at a dose of 240 mg/㎡ was diluted in 500 ml of 5% dextrose solution and infused i.v. for 3 hours on day 1. Specialized i.v. infusion sets or in-line filter was not required for the administration. The dose of Genexol-PM was escalated to 300 mg/㎡ from the second cycle when pre-specified criteria were fulfilled (nadir ANC ≥ 1,000/ mm3, nadir platelet count ≥ 100,000/ mm3, and no grade 2 or worse non-hematologic toxicities with the exception of alopecia)

SUMMARY:
Taxane-based chemotherapy is currently one of the most commonly used regimen for salvage chemotherapy in advanced urothelial carcinoma. In previously untreated patients, single-agent paclitaxel, administered in a 24-hour infusion, produced an overall response rate of 42%, and single-agent docetaxel as a first-line therapy produced response rates of 31% and 45% in 11 patients with impaired renal function. Of the two taxanes, paclitaxel has been studied more extensively.

Intravenous administration of paclitaxel requires the use of solubilizing agents such as Cremophor EL (CrEL) due to its hydrophobicity. CrEL often contributes to hypersensitivity reactions including hypotension or dyspnea with bronchospasm, some of which are major and potentially life-threatening. Minor allergic reactions such as transient rashes and flushing also may occur. Despite pretreatment with corticosteroids and histamine antagonists, minor reactions still occur in 10-44% of all patients, with 1-3% of patients experiencing potentially fatal reactions. CrEL may also act as a potential cofactor for the development of peripheral neuropathy. In addition, special infusion sets must be used clinically when administering CrEL-based paclitaxel.

Genexol-PM (Samyang Co., Seoul, Korea), a form of paclitaxel formulated with sterile, lyophilized polymeric micells that allow intravenous delivery of paclitaxel without CrEL. The polymeric micelle formulation is composed of hundreds of low molecular weight, nontoxic, and biodegradable amphiphilic diblock copolymers which include monomethoxy poly(ethylene glycol)-block-poly(D,L-lactide), and has a great potential in terms of water solubility, in vivo stability, and the nanoscopic size (a diameter of 20-50 nm) of the micellar structure.

A phase I study established that Genexol-PM administered at 390 mg/m2 intravenously for 3 h every 3 weeks was the maximum tolerable dose (MTD) in humans. Dose-limiting toxicities were neuropathy, myalgia, and neutropenia. No hypersensitivity reactions were observed in any patients despite the absence of antiallergic premedication. The recommended dosage for phase II studies was 300 mg/m2.

Based on the promising results of taxane-based chemotherapy and the absence of standard second-line chemotherapy regimen for advanced urothelial cancer, the investigators designed phase II study to explore the efficacy and safety of Genexol-PM in advanced urothelial patients, who previously treated with gemcitabine plus platinum as adjuvant chemotherapy or 1st line therapy for metastatic diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed TCC of the urothelial tract (bladder, renal pelvis, or ureter)
2. Prior exposure to gemcitabine-platinum regimen as either adjuvant or palliative chemotherapy.
3. Unidimensionally measurable disease outside prior radiotherapy ports
4. Age 18 years or older
5. ECOG performance status of 0~2
6. Life expectancy of at least 3 months
7. Adequate BM function (ANC >1,500/mm3 & Platelet >100,000/mm3)
8. Adequate hepatic function (Bilirubin no greater than 2 times upper limit of normal (ULN) & AST or ALT no greater than 2.5 times ULN), and renal function (creatinine <1.5 X times ULN)
9. No pre-existing clinically significant grade 2 or greater neuropathy

Exclusion Criteria:

1. Pregnant or lactating patients
2. Presence or history of CNS metastasis
3. Patients with prior RT to the axial skeleton within 4 weeks of chemotherapy start to greater than 25% of bone marrow
4. Any preexisting medical condition of sufficient severity to prevent full compliance with the study, including active infection, active cardiac symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2007-12; Primary Completion 2010-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Response rate | 6 months
  Objective tumor response rate according to RECIST criteria V.1.0

SECONDARY OUTCOMES:
Adverse events | 12 months
  Adverse events according NCI-CTCAE V3.0
Time to progression | 12 months
  Time from the start of treatment to the objective disease progression
Overall survival | 24 months
  Time from the start of treatment to the date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Lyun Lee, M.D., Ph.D., Study Director — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Result] Lee JL, Ahn JH, Park SH, Lim HY, Kwon JH, Ahn S, Song C, Hong JH, Kim CS, Ahn H. Phase II study of a cremophor-free, polymeric micelle formulation of paclitaxel for patients with advanced urothelial cancer previously treated with gemcitabine and platinum. Invest New Drugs. 2012 Oct;30(5):1984-90. doi: 10.1007/s10637-011-9757-7. Epub 2011 Oct 20. PMID 22012004